CLINICAL TRIAL: NCT01539785
Title: Surgery Plus Hyperthermic Intra-peritoneal Chemotherapy (HIPEC) Versus Surgery Alone in Patients With Platinum-sensitive First Recurrence of Ovarian Cancer: a Prospective Randomized Multicenter Trial.
Brief Title: Hyperthermic Intra-peritoneal Chemotherapy (HIPEC) in Ovarian Cancer Recurrence
Acronym: HORSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Direttore del Dipartimento per la Tutela della salute della Donna e della Vita Nascente Università Cattolica del Sacro Cuore-Roma, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 138/12
Record Dates: First submitted 2012-02-20; First posted 2012-02-28 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: First Recurrence of Ovarian Cancer
Keywords: HIPEC; Hyperthermic; ovarian cancer; recurrence
MeSH Terms: conditions — Fever; Ovarian Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Secondary cytoreduction (Active Comparator): The eligible patients, after anesthesia preparation will be submitted to a surgical complete cytoreduction.
  Interventions: Procedure: Secondary citoreduction
- Hyperthermic intra-peritoneal chemotherapy (HIPEC) (Experimental): If the patient is randomized to make chemo-hyperthermia, surgery will be followed by HIPEC with the closed technique.
  Interventions: Procedure: Hyperthermic intra-peritoneal chemotherapy (HIPEC)

INTERVENTIONS:
Procedure: Secondary citoreduction — The eligible patients, after anesthesia preparation will be submitted to a surgical complete cytoreduction attempt that consist in the removal of all macroscopically visible tumor nodules from the visceral and parietal peritoneum. To obtain a complete cytoreduction, different procedures are required, as described by Sugarbaker (30), which may include omentectomy, splenectomy, diaphragmatic, pelvic,parietal peritonectomy and / or visceral, bowel resection, hepatic resection and cholecystectomy.
  Arms: Secondary cytoreduction
Procedure: Hyperthermic intra-peritoneal chemotherapy (HIPEC) — If the patient is randomized to make chemo-hyperthermia, surgery will be followed by HIPEC with the closed technique, that consist in the perfusion of the abdominal cavity with a solution containing cisplatin (CDDP) 75 mg/m2 in 2L/m2 heated saline. The solution is heated and perfused with two special pumps (Hyperex, Korea or Stoeckert munich). The temperature of inflow and outflow of the solution, will be maintained, respectively, between 41 ° and 42.5 ° C. The intraperitoneal temperature will be maintained at 41.5 ° C and monitored by thermometers inserted into the subphrenic space and into the pelvis. After 60 minutes of perfusion the surgical incision will be open after removal of the entire solution. The global temperature will be measured by thermometer inserted into the esophagus and rectum. A Swan-Ganz catheter will be kept in place during the HIPEC for monitoring cardiovascular function.
  Arms: Hyperthermic intra-peritoneal chemotherapy (HIPEC)

SUMMARY:
The purpose of this study is to determine the role of surgery followed by hyperthermic intra-peritoneal chemotherapy (HIPEC) versus surgery alone in patients with platinum-sensitive first recurrence of ovarian cancer. Moreover it is a prospective randomized multicenter trial, aimed to investigate the prognostic role of surgery plus HIPEC versus surgery alone in terms of progression free interval, overall survival, morbidity and mortality, second recurrence pattern, quality of life with EORTC QLQ-C30 and QLQ OV28 questionnaires.

DETAILED DESCRIPTION:
Among the malignancies of the female genital tract, ovarian cancer is the second most common cancer after the endometrial tumor, but the more lethal, representing the fifth leading cause of death among women in industrialized countries. For the most part, these are epithelial tumors (>70%), who begin with vague gastrointestinal symptoms, general malaise, abdominal bloating, weight loss and fatigue. Because of the non-specificity oh the symptoms and the often late presentation, about 70% of the diagnosis is made at an advanced stage of disease (IIIC). In the last two decades only a modest improvement in survival was achieved. Moreover, even after optimal cytoreduction followed by adjuvant chemotherapy based on platinum and taxane, which is currently the standard for this type of disease, most patients with stage III disease developed a recurrence.

Rational of HIPEC in recurrent ovarian cancer: the cytoreduction. Contrary to what happens in the primary disease is not yet clear what is the standard treatment in recurrent epithelial ovarian cancer (EOC).

Patients who experience a recurrence within 6 months from the end of the first-line chemotherapy are considered platinum-resistant and have applied for a salvage treatment with second line drugs with low response rates and poor survival. Patients who recur after 6 months are considered platinum-sensitive and, therefore, subject to a new chemotherapy treatment with a platinum compound possibly in combination with paclitaxel (re-challenge). In these patients it is possible to achieve a clinical response rate similar to the primary treatment, with median survival reported between 12 and 24 months. Recently surgery affirmed a major role not only in the primary treatment but also in recurrent chemo-sensitive ovarian cancer. A meta-analysis of 2019 patients has shown that obtain an optimal secondary cytoreduction independently correlates with survival (OS) after recurrence. However, a recent Cochrane, showed that, from the studies available nowadays, is not possible to substantiate a difference in prognosis between the exclusive chemotherapy treatment and the association of surgery with adjuvant chemotherapy.

The results of the multicenter trial DESKTOP I show that, even in the presence of peritoneal carcinomatosis, the 2-year survival improves if an optimal cytoreduction is obtained.

Rational of HIPEC in recurrent ovarian cancer: intraperitoneal chemotherapy Many patients who undergo optimal cytoreduction may benefit from adjuvant chemotherapy administered intraperitoneally (IP). Several randomized trials have demonstrated improved survival associated with IP platinum-based chemotherapy as first-line adjuvant therapy after optimal cytoreduction, although it is still unclear which patients might benefit most, or what would be the best drug , its dose or the right number of cycles. The adjuvant IP therapy, however, seems to have more side effects than intravenous therapy (IV) and consequently a worsening of the quality of life (QOL).

Rational use of HIPEC in recurrent ovarian cancer: hyperthermia The association of hyperthermia plus chemotherapy to the surgery based its rational on the cytotoxic effect of hyperthermia, which not only cause a rupture of cell membranes due to protein denaturation (direct effect), but also an increase in the permeability of new vessels and an impairment of receptor protein complexes (indirect effect). The sensitivity of the solid tumors to hyperthermia is probably linked to the creation of a microenvironment with a low pH, low oxygen tension, low glucose levels in response to high temperature. Inactivation of tumor cells is time and temperature dependent, and starts at 40-41 ° C. Experimental data show that human tumor cell lines are more sensitive to a moderate hyperthermia (41-42 ° C).

Furthermore, the ability of its cytotoxic chemotherapeutic agents, including mitomycin C, doxorubicin, cisplatin and oxaliplatin, is enhanced by hyperthermia itself.

Secondary cytoreduction (CRS), HIPEC and ovarian cancer Since its first appearance in 1980, the HIPEC associated with surgery has had an increasingly important role in the treatment of several types of cancer with peritoneal dissemination.

The rational for this therapeutic approach is based on the achievement of higher drug concentrations in contact with the peritoneal surface with a lower systemic concentrations, resulting in a decrease in the systemic toxicity of treatment. The addition of hyperthermia proved to be able to have a cytotoxic effect on tumor cells directly and indirectly, and a synergistic effect with several cytotoxic agents.

Two recent trials including heterogeneous populations of patients with EOC have demonstrated that the use of the HIPEC in association with CRS is followed by an overall survival (OS) of three years after the recurrence that vary between 20-63%. Data from a trial which took place at this Institution and was recently published about the use of HIPEC platinum-sensitive recurrent EOC patients, showed a median disease-free interval (PFS) and OS of 24 and 38 months respectively, with an estimated PFS and OS at 3 years of 44% and 92% respectively. These data not only confirm those previously reported in the literature, but are more significant, probably because of the highly selected population, a characteristic that contrasts with the wide heterogeneity of most of the other trials made until now.

In fact, as demonstrated by the meta-analysis by Bristow et al, the median survival after recurrence in the same group of patients treated with CRS and standard adjuvant chemotherapy alone was 30.3 months. This difference in survival compared with that of our trial could be justified by the increased rate of optimal cytoreduction obtained in our Institution (95.3% vs. 52.2%).

In addition, on the basis of the criteria developed by Markman, that any second-line treatment after recurrence which reaches a PFS similar or comparable to that after the primary disease is considered to be effective, our data show an additional benefit obtained by HIPEC. In the series of patients underwent CRS + HIPEC at this Institution, in fact, the median PFS after primary disease was substantially equal to that after recurrence with values of 25 and 24 months respectively (p = ns). Therefore treatment with CRS associated with HIPEC in with platinum-sensitive recurrent EOC patients would seem to offer the same opportunities in terms of prognosis than primary treatment.

Regarding the complications linked to this procedure, the trials completed at our Institution, showed morbidity and mortality rates about of 35% and 0%, consistent with the data presented by recent review (12 - 52% and 0,9-5,8% respectively), which are however more heterogeneous due to differences between the considered studies. In addition, the analysis divided into two blocks per year of execution of the procedure, has demonstrated a significant reduction in the percentage of complications (up to 26.7%) with a statistically significant difference.

Currently, despite the presence of a strong biological and pharmacological rational and the over 10 years application in EOC, the use of HIPEC in the clinical practice continues to receive mixed reviews. The limit to the confidence in this procedure is the lack of randomized clinical trials and the heterogeneity of the different phase II studies conducted, which resulted in a lack of scientific evidence level I-II. Moreover, the finding of high rates of the related morbidity and mortality, has precluded the use of this procedure to many patients with peritoneal disease.

The primary objective of this trial is therefore to assess whether the use of CRS in combination with HIPEC is able to offer an effectively advantage in terms of survival compared to the exclusive optimal CRS, in platinum-sensitive recurrent EOC patients, whom potentially could undergo complete cytoreduction on the basis of the pre-and intraoperative evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 and under 70 years
* Patients affected by a first recurrence of ovarian cancer with measurable lesions or not, but evaluable (upwards of Ca125 for 2 consecutive assessments).
* ECOG-performance status ≤ 2
* Ovarian cancer limited to the abdominal cavity with or without extraperitoneal spread considered resectable at intraoperative evaluation
* Evidence of tumor recurrence diagnosed after 6 months from primary treatment
* Previous-based chemotherapy of carboplatin and taxanes
* Positive Peritoneal Washing in the presence of other abdominal disease surgically resectable
* Adequate respiratory, hepatic, cardiac, kidney and bone marrow function (absolute neutrophil count > 1500/mm3, platelets > 150,000/μl, creatinine clearance > 60 mL/min according to Cockroft formula)
* Patient-compliant and psychologically able to follow the trial procedures

Exclusion Criteria:

* Non-epithelial ovarian cancer or borderline ovarian tumor
* Pregnancy or breastfeeding
* Patients affected by major depressive disorder even in treatment or minor mood disorders
* Patients with severe impairment of respiratory, hepatic or renal function
* Patients with cardiac, neurological or metabolic uncontrolled pharmacologically disease
* Patients with active infection or other neoplastic disease in progress
* Patients with bowel obstruction
* Inadequate bone marrow, liver, kidney function
* No clear-peritoneal disease at surgical exploration
* Patients with ascites > 500 ml (the TAC)
* Patients on maintenance therapy with Antiangiogenic drugs
* Patients with secondary or tertiary recurrence, or already submitted to HIPEC
* Patients who have already made the second or third line chemotherapy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Estimate of progression free interval (PFI) in the two trial arms. | 36 months
  The progression-free interval (PFI) will be evaluated from the time of secondary cytoreduction (± HIPEC) to the evidence of a second recurrence of disease.

SECONDARY OUTCOMES:
Estimate of overall survival (OS)in the two trial arms. | 36 months
  The overall survival (OS) will be evaluated from the time of secondary cytoreduction ± HIPEC to death or last FU.
Evaluation of the morbidity and mortality in the two trial arms. | 36 months
  Surgical complications and morbidity will be monitored and recorded in special forms both during surgery and during the period of hospital stay. The following complications should be reported to the coordinating center UCSC within 24 hours Events recorded during surgery and up to 60 days of the latter: transfusion of more than 10 units of blood in 24 hours, re-laparotomy for complications, pulmonary embolism, sepsis, death (regardless of cause), new hospitalization for surgical complication.
  Events between 60 days and the end of follow-up period: death (regardless of cause).

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred the Hearth, Rome, Rome, Italy

REFERENCES:
- [Derived] Fagotti A, Costantini B, Fanfani F, Giannarelli D, De Iaco P, Chiantera V, Mandato V, Giorda G, Aletti G, Greggi S, Perrone AM, Salutari V, Trozzi R, Scambia G. Hyperthermic Intraperitoneal Chemotherapy in Platinum-Sensitive Recurrent Ovarian Cancer: A Randomized Trial on Survival Evaluation (HORSE; MITO-18). J Clin Oncol. 2025 Mar;43(7):852-860. doi: 10.1200/JCO.24.00686. Epub 2024 Nov 21. PMID 39571127
- [Derived] Petrillo M, Zucchetti M, Cianci S, Morosi L, Ronsini C, Colombo A, D'Incalci M, Scambia G, Fagotti A. Pharmacokinetics of cisplatin during open and minimally-invasive secondary cytoreductive surgery plus HIPEC in women with platinum-sensitive recurrent ovarian cancer: a prospective study. J Gynecol Oncol. 2019 Jul;30(4):e59. doi: 10.3802/jgo.2019.30.e59. Epub 2019 Mar 1. PMID 31074245
- [Derived] Fagotti A, Petrillo M, Costantini B, Fanfani F, Gallotta V, Chiantera V, Turco LC, Bottoni C, Scambia G. Minimally invasive secondary cytoreduction plus HIPEC for recurrent ovarian cancer: a case series. Gynecol Oncol. 2014 Feb;132(2):303-6. doi: 10.1016/j.ygyno.2013.12.028. Epub 2013 Dec 27. PMID 24378877